CLINICAL TRIAL: NCT02955615
Title: A Phase II, Multi-centre, Randomized, Double Blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Pharmacokinetics of ILT-101 in Patients With Active Moderate to Severe Systemic Lupus Erythematosus (SLE)
Brief Title: ILT-101 in Patients With Active Moderate to Severe Systemic Lupus Erythematosus (SLE)
Acronym: LUPIL-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iltoo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-002; 2016-000488-17 (EudraCT Number)
Record Dates: First submitted 2016-10-17; First posted 2016-11-04 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ILT-101 (Experimental): Subcutaneous administrations for 3 to 6 months according to clinical responder status at week 12
  Interventions: Drug: ILT-101
- Placebo (Placebo Comparator): Subcutaneous administrations for 3 to 6 months according to clinical responder status at week 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ILT-101 — Induction phase followed by weekly administrations of ILT-101 on top of SLE background therapy.
  SLE background therapy includes ...
  Other Names: Low dose IL-2
  Arms: ILT-101
Drug: Placebo — Induction phase followed by weekly administrations of placebo on top of SLE background therapy.
  SLE background therapy includes ...
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ILT-101 (human recombinant interleukin 2 (IL-2)) in patients with moderate to severe systemic lupus erythematosus.

DETAILED DESCRIPTION:
Interleukin 2 (IL-2) plays an important role on immune homeostasis by acting on T lymphocytes. In systemic lupus erythematosus, there is a so called "insufficiency" in a subpopulation of T lymphocytes, the regulatory T cells (Tregs) leading to altered immune balance between regulatory and effector T cells. These cells seem to play a major role in the physiopathology of the disease. Many researches enlighten the fact that this Tregs/Teffs balance can be restored by administering low dose of IL-2. It is thus assumed that treatment with low dose of IL-2 may impact positively the progression of the disease and thus help patients improving their clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SLE
* Active SLE
* On stable background therapy for 1 month
* Using highly effective contraception

Exclusion Criteria:

* Serious organ failure (renal functional impairment, severe central nervous system manifestations, severe heart failure, liver failure)
* Any clinical evidence of active chronic infection HIV, hepatitis B, hepatitis C
* Clinical significant pleuritis or pericarditis
* Type1 Diabetes and/or CROHN's disease
* Use of Benlysta (belimumab) in the past 4 weeks
* Use of Rituximab in the past 6 months
* Vaccination with live attenuated virus in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
SRI-4 (SLE responder index) | at week 12
  Number of participants with SRI-4

SECONDARY OUTCOMES:
Incidence of adverse events | From baseline up to week 24 or 36
Number of participants able to reduce oral steroid dose of 25 and 50% | From baseline to week 12 or 24
Anti ds-DNA by immunology-based assay | From baseline to week 12 or 24
  Change in anti-dsDNA as compared to baseline
%Tregs | From baseline to week 12 or 24
  % change in Tregs as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: David Klatzmann, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris (AP-HP)
Locations (25):
- AKH Wien, Vienna, Austria
- Bulgaria (2):
  - University Multiprofile Hospital for Active Treatment, Plovdiv
  - University Multiprofile Hospital, Sofia
- France (3):
  - Hopital Claude Huriez, Lille
  - Hopital Européen, Marseille
  - Hôpital Haut Lévèque, Pessac
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt am Main
  - University Clinic Leipzig AöR, Leipzig
  - University Clinic Schleswig-Holstein, Lübeck
- Azienda Osp. Univ. Seconda Università di Napoli, Napoli, Italy
- Cap research, Phoenix, Mauritius
- Mexico (5):
  - Hospital AmeriMed Cons., Cancún
  - Investigación y Biomedicina, Chihuahua City
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Centro Integral en Reumatología S.A. de C.V., Guadalajara
  - Clitider S.A. de C.V., Mexico City
- Portugal (2):
  - Hospital Prof. Doutor Fernando Fonseca, Amadora
  - Centro Hospitalar de Lisboa Ocidental, Lisbon
- Romania (3):
  - Neomed, Brasov
  - Euroclinic Hospital, Bucharest
  - Sf. Maria Hospital, Bucharest
- Spain (3):
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Humrich JY, Cacoub P, Rosenzwajg M, Pitoiset F, Pham HP, Guidoux J, Leroux D, Vazquez T, Riemekasten G, Smolen JS, Tsokos G, Klatzmann D. Low-dose interleukin-2 therapy in active systemic lupus erythematosus (LUPIL-2): a multicentre, double-blind, randomised and placebo-controlled phase II trial. Ann Rheum Dis. 2022 Dec;81(12):1685-1694. doi: 10.1136/ard-2022-222501. Epub 2022 Aug 16. PMID 35973803